CLINICAL TRIAL: NCT05002998
Title: A Phase 3b/4, Double-masked, Randomized, International, Parallel-assignment, Multicenter Trial in Patients With Thyroid Eye Disease to Evaluate the Safety and Tolerability of Different Dosing Durations of Teprotumumab
Brief Title: TEPEZZA® (Teprotumumab-trbw) Post-Marketing Requirement Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HZNP-TEP-402; 2020-005999-36 (EudraCT Number); 2024-515090-96-00 (EU CTIS Number)
Record Dates: First submitted 2021-07-19; First posted 2021-08-12 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Thyroid Eye Disease
Keywords: TED
MeSH Terms: conditions — Graves Ophthalmopathy | interventions — teprotumumab; Saline Solution

STUDY DESIGN:
Intervention Model Description: * 4 infusions of teprotumumab (10 mg/kg for the first infusion and 20 mg/kg for the remaining 3 infusions) (Cohort 1) followed by 4 infusions of:
    * Placebo if a participant is a treatment responder at Week 12 or
    * Teprotumumab 20 mg/kg if a participant is a treatment non-responder at Week 12
  * 8 infusions of teprotumumab (10 mg/kg for the first infusion and 20 mg/kg for the remaining 7 infusions) (Cohort 2)
  * 16 infusions of teprotumumab (10 mg/kg for the first infusion and 20 mg/kg for the remaining 15 infusions) (Cohort 3)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-masked except for the pharmacy staff.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Teprotumumab 4 Infusions (Other): • 4 infusions of teprotumumab (10 mg/kg for the first infusion and 20 mg/kg for the remaining 3 infusions) (Cohort 1) followed by 4 infusions of:
  * Placebo if a participant is a treatment responder at Week 12 or
  * Teprotumumab 20 mg/kg if a participant is a treatment non-responder at Week 12
  Interventions: Drug: Teprotumumab; Drug: Placebo
- Teprotumumab 8 Infusions (Other): 8 infusions of teprotumumab (10 mg/kg for the first infusion and 20 mg/kg for the remaining 7 infusions) (Cohort 2)
  Interventions: Drug: Teprotumumab
- Teprotumumab 16 Infusions (Other): 16 infusions of teprotumumab (10 mg/kg for the first infusion and 20 mg/kg for the remaining 15 infusions) (Cohort 3)
  Interventions: Drug: Teprotumumab

INTERVENTIONS:
Drug: Teprotumumab — Teprotumumab is a fully human anti-IGF-1R mAb. Teprotumumab will be provided in single-dose 20-mL glass vials as a freeze-dried powder containing, in addition to the drug substance, 20 mmol/L histidine-histidine chloride, 250 mmol/L trehalose and 0.01% polysorbate 20 (w/w).
  Prior to administration, each vial containing 500 mg teprotumumab freeze-dried powder will be reconstituted with 10 mL of sterile water for injection. The resulting solution will have a concentration of 47.6 mg/mL teprotumumab-trbw antibody. The reconstituted teprotumumab solution must be further diluted in 0.9% (w/v) sodium chloride (NaCl) solution prior to administration
  Other Names: TEPEZZA
Drug: Placebo — Placebo will consist of a normal saline (0.9% NaCl) solution and will be administered in 100 mL or 250 mL infusion bags, as appropriate, per weight-based dosing volumes.
  Other Names: Saline Solution
  Arms: Teprotumumab 4 Infusions

SUMMARY:
This is a double-masked, randomized, parallel-assignment, multicenter trial examining the safety and tolerability of teprotumumab in the treatment of Thyroid Eye Disease (TED) in adult participants. This international, Phase 3b/4 trial is being conducted to fulfill an FDA post-marketing requirement for a descriptive trial to evaluate the safety, efficacy and need for re-treatment of 3 different teprotumumab treatment durations for TED. In addition, serum samples from participants with a Baseline Clinical Activity Score (CAS) ≥3 will be evaluated for biomarkers of disease.

DETAILED DESCRIPTION:
Participants will be screened for eligibility within 4 weeks prior to the Baseline (Day 1) Visit. Approximately 300 participants who meet the trial eligibility criteria will be randomized on Day 1 in a 1:1:1 ratio in a double-masked fashion (stratified by CAS(clinical activity score) [≥3 (active) or <3 (inactive)] and disease severity [severe disease, defined as both proptosis above normal for race and gender with binocular diplopia at Baseline vs. non-severe disease]) to receive:

* 4 infusions of teprotumumab (10 mg/kg for the first infusion and 20 mg/kg for the remaining 3 infusions) (Cohort 1) followed by 4 infusions of:

  * Placebo if a participants is a treatment responder at Week 12 or
  * Teprotumumab 20 mg/kg if a participant is a treatment non-responder at Week 12
* 8 infusions of teprotumumab (10 mg/kg for the first infusion and 20 mg/kg for the remaining 7 infusions) (Cohort 2)
* 16 infusions of teprotumumab (10 mg/kg for the first infusion and 20 mg/kg for the remaining 15 infusions) (Cohort 3)

Three weeks following the final infusion of the Initial Treatment Period, there will be a comprehensive End-of-Initial Treatment Visit at Week 24 (Cohorts 1 and 2)/Week 48 (Cohort 3). At this visit, all participants will be assessed for treatment response.

Proptosis responders in all cohorts and non-responders in Cohorts 1 and 2 who choose not to receive a second treatment course, will enter a 52 week Initial Follow-up Period.

Proptosis non-responders in Cohorts 1 and 2 who choose to receive a second treatment course (8 infusions) of teprotumumab will receive an infusion q3W.

Proptosis non-responders in Cohort 3 are not eligible for a second treatment course following initial treatment.

Participants in any of the 3 cohorts who are proptosis responders following the Initial Treatment Period and who flare during the Initial Follow up Period will be eligible to receive re treatment.

Acquired from Horizon in 2024

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent.
2. Male or female between the ages of 18 and 80 years, inclusive, at Screening.
3. Initial diagnosis of TED within 7 years prior to Screening.
4. Proptosis ≥3 mm from baseline (prior to diagnosis of TED), as estimated by treating physician, and/or proptosis >3 mm above normal for race and gender.
5. Participants must be euthyroid with the baseline disease under control or have mild hypo or hyperthyroidism (defined as free thyroxine and free triiodothyronine levels <50% above or below the normal limits) at Screening. Every effort should be made to correct the mild hypo- or hyperthyroidism promptly and to maintain the euthyroid state for the duration of the trial.
6. Does not require immediate surgical ophthalmological intervention and is not planning corrective surgery/irradiation during the course of the trial.
7. Diabetic participants must have HbA1c ≤8.0% at Screening.
8. Participants with a history of IBD (ulcerative colitis or Crohn's disease) must be in clinical remission for at least 3 months, with no history of bowel surgery within 6 months prior to Screening and no planned surgery during the trial. Concomitant stable therapies for IBD without modifications in the 3 months prior to Screening are allowed.
9. Women of childbearing potential (including those with an onset of menopause <2 years prior to Screening, non-therapy-induced amenorrhea for <12 months prior to Screening or not surgically sterile [absence of ovaries and/or uterus]) must have a negative serum pregnancy test at Screening and negative urine pregnancy tests at all protocol-specified time points (i.e., prior to each dose and throughout the participant's participation in the Follow-up Period); participants who are sexually active with a non-vasectomized male partner must agree to use 2 reliable forms of contraception during the trial, 1 of which is recommended to be hormonal, such as an oral contraceptive. Hormonal contraception must be started at least 1 full cycle prior to Baseline and continue for 180 days after the last dose of teprotumumab. Highly effective contraceptive methods (with a failure rate <1% per year), when used consistently and correctly, include implants, injectables, combination oral contraceptives, some intrauterine devices, tubal ligation, sexual abstinence or vasectomized partner.
10. Willing and able to comply with the prescribed treatment protocol and evaluations for the duration of the trial.

Exclusion Criteria:

1. Decreased best-corrected visual acuity due to optic neuropathy, as defined by a decrease in vision of 2 lines on the Snellen chart, new visual field defect or color defect secondary to optic nerve involvement within the last 6 months.
2. Corneal decompensation unresponsive to medical management.
3. Decrease in proptosis of ≥2 mm in the study eye between Screening and Baseline.
4. Prior orbital irradiation, orbital decompression or strabismus surgery.
5. Planned eyelid surgery during the course of the trial.
6. Alanine aminotransferase or aspartate aminotransferase >3 × the upper limit of normal or estimated glomerular filtration rate ≤30 mL/min/1.73m2 at Screening.
7. Use of any steroid (intravenous [IV], oral, steroid eye drops) for the treatment of TED or other conditions within 3 weeks prior to Screening. Steroids cannot be initiated during the trial. Exceptions include topical and inhaled steroids, as well as steroids used to treat infusion reactions.
8. Any treatment with rituximab (Rituxan® or MabThera®) within 12 months prior to the first infusion of teprotumumab or tocilizumab (Actemra® or Roactemra®) within 6 months prior to the first infusion of teprotumumab. Use of any other non-steroid immunosuppressive agent within 3 months prior to the first infusion of teprotumumab.
9. Any previous treatment with teprotumumab, including previous enrollment in this trial or participation in a prior teprotumumab trial.
10. Treatment with any mAb within 3 months prior to Screening.
11. Identified pre-existing ophthalmic disease that, in the judgment of the Investigator, would preclude trial participation or complicate interpretation of trial results.
12. Use of an investigational agent for any condition within 60 days or 5 half-lives, whichever is longer, prior to Screening or anticipated use during the course of the trial.
13. Malignant condition in the past 5 years (except successfully treated basal/squamous cell carcinoma of the skin or cervical cancer in situ).
14. Pregnant or lactating women.
15. Current drug or alcohol abuse or history of either within the previous 2 years, in the opinion of the Investigator or as reported by the participant.
16. Known hypersensitivity to any of the components of teprotumumab or prior hypersensitivity reactions to mAbs.
17. Human immunodeficiency virus, untreated or positive viral load for hepatitis C or hepatitis B infections.
18. Any other condition that, in the opinion of the Investigator, would preclude inclusion in the trial.
19. After 150 participants with a CAS <3 at Baseline have been randomized, an additional exclusion criterion will apply: CAS <3 at Baseline.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 313 (Actual)
Dates: Start 2021-09-16 (Actual); Primary Completion 2025-12-19 (Actual); Study Completion 2025-12-19 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants who experience at least 1 treatment-emergent adverse event (TEAE) and the percentage of participants who experience at least 1 treatment emergent AESI during treatment with teprotumumab | Screening to End of Study (last visit possible is Week 136)
  Treatment emergent adverse events and treatment emergent adverse events of special interest will be evaluated from the beginning of the study until follow up.
Percentage of Participants who receive re-treatment | Week 27 to Week 136
  Participants who are not proptosis responders after initial treatment or participants who are proptosis responders after initial treatment but who have flared during follow-up (relapsed).

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (28):
- United States (7):
  - The Private Practice of Raymond Douglas, MD - Beverly Hills, Beverly Hills, California
  - USC Roski Eye Institute - Los Angeles, Los Angeles, California
  - Stanford University, Palo Alto, California
  - University of Colorado - Eye Center - PPDS, Aurora, Colorado
  - Bascom Palmer Eye Institute, Miami, Florida
  - Mayo Clinic - PPDS, Rochester, Minnesota
  - Casey Eye Institute - OHSU, Portland, Oregon
- France (4):
  - Hopital Jean Minjoz, Besançon, Doubs
  - Hospices Civils de Lyon - Hôpital Louis Pradel, Bron, Rhône
  - Hôpital Claude Huriez-Lille-Rue Michel Polonovski, Lille
  - Centre Hospitalier National D'ophtalmologie Des Quinze Vingts, Paris
- Germany (5):
  - Universitätsklinikum Tübingen, Tübingen, Baden-Wurttemberg
  - University Medicine Göttingen Germany, Göttingen, Lower Saxony
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz, Rhineland-Palatinate
  - Universitätsklinikum Essen, Essen
  - Universitätsklinikum Münster, Münster
- Italy (4):
  - Azienda Ospedaliera Universitaria Federico II, Napoli, Campania
  - ASST dei Sette Laghi - Ospedale Di Circolo E Fondazione Macchi, Varese, Lombardy
  - ARNAS Garibaldi - PO Garibaldi-Centro, Catania, Sicily
  - Azienda Ospedaliero Universitaria Pisana - Stabilimento Santa Chiara, Pisa, Tuscany
- Spain (3):
  - Hospital La Arruzafa, Córdoba, Córdoba
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario Virgen Macarena, Seville
- United Kingdom (5):
  - Moorfields Eye Hospital - PPDS, London, London, City of
  - Imperial College Healthcare NHS Trust - PPDS, London, London, City of
  - University Hospital of Cardiff, Cardiff, South Glamorgan
  - Royal Victoria Infirmary, Newcastle upon Tyne, Tyne and Wear
  - Southampton University Hospitals NHS Trust, Southampton

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Related Info — http://www.TEPEZZA.com